CLINICAL TRIAL: NCT03054740
Title: Will Patients Perceive a Vapocoolant Spray to be Effective in Reducing Pain and Increasing Satisfaction With Insertion at an Intravenous Site?
Brief Title: Vapocoolant Spray Used Prior to Intravenous (IV) Insertions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AultmanHF
Record Dates: First submitted 2017-02-06; First posted 2017-02-16 (Actual); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Pain
Keywords: Vapocoolant applied prior to IV access
MeSH Terms: conditions — Pain | interventions — Ethyl Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gebauer Ethyl Chloride (Active Comparator): Device: Vapocoolant (Ethyl Chloride Mist Spray)
  Interventions: Drug: Gebauer Ethyl Chloride
- Nature's Tears (Placebo Comparator): Device: Sterile Water
  Interventions: Drug: Nature's Tears

INTERVENTIONS:
Drug: Gebauer Ethyl Chloride — Will be administered according to manufacturers recommendations which is to spray the aerosol can for 4-10 seconds from a distance of 3 to 9 inches. Do not spray longer than 10 seconds.
  Other Names: Ethyl Chloride Mist Spray Can
  Arms: Gebauer Ethyl Chloride
Drug: Nature's Tears — Sterile water mist will be administered 1-2 sprays prior to intravenous access
  Other Names: Sterile Water
  Arms: Nature's Tears

SUMMARY:
The primary purpose of this study is to determine if by offering a vapocoolant (cold spray) to hospital outpatients prior to an intravenous catheter (IV) insertion will increase patient satisfaction of IV insertion as well as determine if pain of insertion is decreased.

DETAILED DESCRIPTION:
This is a single blind interventional study with a post design using a convenience sample of patients undergoing a Nuclear Medicine Stress Test. The patient selection and intervention will be randomized in order to ensure a high validity study. The interventional treatment used will be a ethyl chloride mist spray manufactured by the Gebauer Company. The placebo spray that will be used is manufactured by BioLogic Aqua Research Technologies International Inc. The spray is called Nature's Tears Mist and is a sterile water. The patient's for this study are required to have intravenous cannulation (IV) access. This is a painful and invasive procedure in which a vapocoolant may confer benefit for the relief of pain.

ELIGIBILITY:
Inclusion Criteria:

* Any outpatient ordered to undergo a Nuclear Medicine Stress Test and is required to have IV access for injection of Radiopharmaceuticals

Exclusion Criteria:

* If it is the first time the patient has had an intravenous catheter inserted
* Any patient who is or may be pregnant
* Any patient who is breast-feeding
* Any patient who has taken a narcotic, sedative and/or anti-anxiety medication within 8 hours of intervention time.
* Any patient who has a known diagnosis of Raynaud's Syndrome or Carpal Tunnel Syndrome.
* Any patient who has an allergy or hypersensitivity to Ethyl Chloride.
* Any patient under the age of 18 and/or any patient over the age of 85
* Any patient who is illiterate
* Any patient who is non-English speaking
* Any patient with prior experience with a vapocoolant spray.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitryn Kar, M.D., Principal Investigator — Aultman Hospital- Interventional Radiologist
Locations (1):
- Aultman Health Foundation, Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffith RJ, Jordan V, Herd D, Reed PW, Dalziel SR. Vapocoolants (cold spray) for pain treatment during intravenous cannulation. Cochrane Database Syst Rev. 2016 Apr 26;4(4):CD009484. doi: 10.1002/14651858.CD009484.pub2. PMID 27113639
- [Background] Levitt FC, Ziemba-Davis M. An exploratory study of patient preferences for pain management during intravenous insertion: maybe we should sweat the small stuff. J Perianesth Nurs. 2013 Aug;28(4):223-32. doi: 10.1016/j.jopan.2012.11.008. PMID 23886287
- [Background] Mace SE. Prospective, randomized, double-blind controlled trial comparing vapocoolant spray vs placebo spray in adults undergoing venipuncture. Am J Emerg Med. 2016 May;34(5):798-804. doi: 10.1016/j.ajem.2016.01.002. Epub 2016 Jan 7. PMID 26979261

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gebauer Ethyl Chloride | Nature's Tears
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gebauer Ethyl Chloride | Nature's Tears | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 8 | 20
  >=65 years | 3 | 7 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Scale Using Visual Analog Scale
Description: 0-No Pain; 1-3 Mild Pain; 4-6 Moderate-Severe Pain; 7-9 Very Severe Pain;10 Worst Possible Pain
Time Frame: less than 5 minutes following spray application
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gebauer Ethyl Chloride | Nature's Tears
Number analyzed (Participants) | 15 | 15
score on a scale | 1.13 (1.302) | 1.60 (1.639)
Statistical Analysis 1: Comparison: Gebauer Ethyl Chloride vs Nature's Tears; Test type: Superiority; Levene's Test of Equality of Error Variances (Design: Intercept + Pain Previous IV + Intervention) F = .001, df1 = 1, df2=28, Sig. = .972

2. Secondary Outcome: Satisfaction Scale Using 1-5 Likert Scale
Description: 1-Very Satisfied; 2-Somewhat Satisfied; 3-Neither Satisfied or Dissatisfied; 4-Somewhat Satisfied; 5-Very Satisfied
Time Frame: less than 5 minutes following spray application
Measure: Count of Participants; unit: Participants
Arm/Group | Gebauer Ethyl Chloride | Nature's Tears
Number analyzed (Participants) | 15 | 15
Participants
  Somewhat Satisfied | 2 | 5
  Very Satisified | 13 | 10
Statistical Analysis 1: Comparison: Gebauer Ethyl Chloride vs Nature's Tears; Test type: Superiority; p = .390, Fisher Exact

3. Secondary Outcome: Using the Same Likert Scale Rate How Satisfied the Patient Remembers the Last Time They Had IV Catheter Inserted
Description: 1-5 Likert Scale
  1 very dissatisfied, 2 somewhat dissatisfied, 3 neither satisfied or dissatisfied, 4 somewhat satisfied, 5 very satisfied
Time Frame: At baseline prior to spray application
Measure: Count of Participants; unit: Participants
Arm/Group | Gebauer Ethyl Chloride | Nature's Tears
Number analyzed (Participants) | 15 | 15
Participants
  Very Dissatisified | 1 | 0
  Somewhat Dissatisfied | 2 | 1
  Neither Satisified or Dissatisfied | 0 | 1
  Somewhat Satisfied | 10 | 12
  Very Satisfied | 2 | 1

4. Secondary Outcome: Using the Same Visual Analog Scale Rate Pain the Last Time the Patient Remembers Having an IV Inserted
Description: Visual Analog Scale 0 no pain, 1-2 mild, 3-5 moderate, 6 severe, 7-8 very severe, 9-10 worst possible pain
Time Frame: At baseline prior to spray application
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gebauer Ethyl Chloride | Nature's Tears
Number analyzed (Participants) | 15 | 15
score on a scale | 3.40 (2.746) | 2.87 (2.031)

5. Secondary Outcome: Would Patient Choose to Have Intervention Again if IV Catheter Insertion is Needed
Description: Yes or No question
Time Frame: less than 10 minutes following spray application
Measure: Count of Participants; unit: Participants
Arm/Group | Gebauer Ethyl Chloride | Nature's Tears
Number analyzed (Participants) | 15 | 15
Participants
  Yes | 12 | 8
  No | 3 | 7

ADVERSE EVENTS:
Time Frame: 2 hours
Groups:
- Gebauer Ethyl Chloride: Drug: Vapocoolant (Ethyl Chloride Mist Spray)
  Gebauer Ethyl Chloride: Will be administered according to manufacturers recommendations which is to spray the aerosol can for 4-10 seconds from a distance of 3 to 9 inches. Do not spray longer than 10 seconds.
- Nature's Tears: Drug: Sterile Water
  Nature's Tears: Sterile water mist will be administered 1-2 sprays prior to intravenous access
Arm/Group | Gebauer Ethyl Chloride | Nature's Tears
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT03054740/Prot_SAP_000.pdf